CLINICAL TRIAL: NCT06023628
Title: Characteristics of Patients With Traumatic Cardiac Arrest in Denmark Assessed by the Danish Helicopter Emergency Medical Services
Brief Title: Patients With Traumatic Cardiac Arrest Assessed by the Danish HEMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Signe Amalie Wolthers, Principal investigator, Prehospital Center, Region Zealand
Other Study IDs: TCA_HEMS_2023
Record Dates: First submitted 2023-03-05; First posted 2023-09-05 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Trauma
Keywords: Traumatic cardiac arrest; Emergency medical services
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Danish Helicopter Emergency Service — Patients with traumatic cardiac arrest assessed by the Danish HEMS

SUMMARY:
This study evaluates patients suffering from traumatic cardiac arrest assessed by the Danish HEMS between 2016 and 2021. The primary outcome is 30-day survival; secondary outcomes are status at admission to the hospital and prehospital return of spontaneous circulation. Further, the prehospital critical care was identified and evaluated.

DETAILED DESCRIPTION:
Background Traumatic cardiac arrest (TCA) is associated with a poor prognosis, [1-3] and prompt, evidence-based treatment is paramount for increasing survival rates.

Cardiac arrest from traumatic origin is characterised as the end state of decompensated haemorrhagic shock, hypoxemia and/or obstructive shock.[1,4] Hypovolaemia and traumatic brain injury account for most cases, accounting for almost 90% of all TCAs.[5] Managing TCA relies on a time-critical assessment of reversible causes, which takes priority over chest compressions and simultaneous management of reversible causes.[1] Thus, TCA mandates urgent action in specialised prehospital treatment and further in-hospital advanced care in specialised trauma centres. [1] Potentially reversible causes of TCA include hypoxaemia, hypovolaemia and obstructive shock.[1,4] Earlier, resuscitation from TCA was considered futile due to meagre survival rates, yet survival has improved through the last decades. [5] Still, substantial variations in survival are seen across different populations. [4-7] Rapid transportation to specialised capacity, the role of the HEMS as an integrated function of the trauma system and the expertise of the helicopter crew are all factors that have been used to explain the benefits associated with using the HEMS in the trauma setting. [8-10] In-depth knowledge of the epidemiology of TCA is essential to improve care within this diverse subgroup of cardiac arrests. The hypothesis is that this novel data on TCA provide new and central data on reversible causes and treatment of these, which are linked to enhanced survival of cardiac arrest of traumatic origin.

Thus, the primary objective of the present study is to investigate the characteristics of patients to whom the Danish HEMS was dispatched who suffered from TCA. This assessment will be done by assessing the incidence, prognostic factors, critical care interventions, and survival from cardiac arrest of traumatic origin.

Materials and Methods This retrospective population-based cohort study with 30-day follow-up includes data from the national HEMS database on patients with traumatic cardiac arrest between 2014 and 2022. Patients will be included if the HEMS physician clinically assessed them and diagnosed them with OHCA from traumatic origin. Hence, patients declared dead on scene by the HEMS will be included. The traumatic aetiology will be supported by secondary diagnoses and free text descriptions from the HEMS database. Trigger words are developed using consecutive text search algorithms in a predefined subgroup of all OHCAs in the Danish Cardiac Arrest Registry note fields. The text search algorithm has been manually validated until no further relevant cases came up.

Data acquisition The HEMS file data were linked to the Danish Civil Registration System and, finally, to the prehospital patient record through the personal civil identification number. The HEMS file database was established in October 2014 and comprises information on all HEMS dispatches in Denmark.[12] Variables included

* Age: Age will be defined as the subject age at the time of the event.
* Sex: Sex will be defined as either male, female or undetermined and derived from the personal civil identification number
* Initial rhythm: The initial rhythm will be defined as the first rhythm observed by the first EMS personnel at the scene. The initial rhythm will be categorised as shockable, non-shockable (asystole), non-shockable (other) or undetermined. In case of conflicting data, the initial rhythm reported by the physician will be used. The initial rhythm will be derived from the prehospital patient record or the HEMS file text.
* Location of Incidence: The location will be either a residential area, outdoors and nature, private home or other. The location will be derived from the prehospital patient record and the HEMS file text.
* Observation of occurrence: Cardiac arrests will be defined as unwitnessed, bystander witnessed or EMS-witnessed. The observation of occurrence will be derived from the prehospital patient record and the HEMS file text.
* Mechanism of injury: Will be classified as blunt (high or low level of energy), penetrating or burn injury, according to the Utstein template. [13]
* Classification of trauma: Will be classified as road collisions, falls from less than two metres, falls from more than two metres, blunt trauma (miscellaneous), gunshot wounds, sharp force trauma, and burns.
* Cardio-pulmonary-resuscitation (CPR): CPR will include bystander-initiated CPR and EMS treatment with CPR. The presence of CPR will be derived from the prehospital patient record and the HEMS file text.
* Defibrillation and use automatic external defibrillators (AEDs): Defibrillation will include defibrillation by bystanders and EMS personnel. Use of AEDs includes using the device if it does not deliver shocks. The status of defibrillation or use of an AED will be derived from the prehospital patient record and the HEMS file text.
* Response time: This will be defined as the time between a dispatcher receiving the emergency call and the arrival of the first EMS personnel. Response time for arrival of the HEMS will be stated as well.
* Time on the scene: Time on the scene is defined as the time between the arrival of the first EMS personnel and departure of the HEMS/ambulance or in case of termination of treatment.
* Hospitalisation: Hospitalisation will be considered either transported to the hospital or declared dead by EMS personnel.
* Prehospital Return-of-spontaneous-circulation (ROSC): ROSC will be classified as the achievement of ROSC anytime between recognition of the event and termination (defined as either hospital admission or declaration of death by EMS personnel).
* State at hospital admission: The state of the case upon arrival at the hospital will be defined as either ROSC or ongoing CPR.
* Survival: 30-day survival, derived from Danish Civil Registration System data.
* Airway management: This includes the airway manoeuvres performed in each case. It is defined by listing the use of airway adjuncts such as nasopharyngeal airway, oropharyngeal airway, endotracheal intubation, supraglottic airway device, and isolated bag-valve-mask ventilation. The airway management will be derived from the prehospital patient record and the HEMS file.
* Automated chest compressions: Use of automated chest compression device. The use of mechanical chest compression devices will be derived from the prehospital patient record and the HEMS file
* Ultrasound examination: Any ultrasound examination of patients. The use of ultrasound will be derived from the prehospital patient record and the HEMS file
* Pleural drainage: This includes chest tube insertion and thoracotomy. The presence of pleural drainage will be derived from the prehospital patient record and the HEMS file
* Blood products: Prehospital transfusion with blood products.
* Prehospital medication: Medication such as tranexamic acid, adrenalin, and calcium will be a binary variable. It is derived from the prehospital patient record and the HEMS file text.
* Other prehospital treatment/management: Use of Tourniquets, the performance of clam-shell thoracotomy, iTClamp (Innovative Trauma Care, San Antonio, TX, USA)

Participants This study includes all patients with TCA in Denmark between 2016 and 2021 who were treated by the Danish HEMS. All age groups are included. Patients will be included if they suffered from an OHCA from traumatic origin and were assessed by the Danish HEMS. The latter will be identified through manual validation based on a predefined search string among all OHCAs in Denmark (derived from the Danish Cardiac Arrest Registry) within the study period. TCA is defined as cardiac arrest resulting from blunt, penetrating or burn injury, according to the Utstein template.[11] Patients to whom the HEMS was dispatched but did not arrive will be excluded. Patients with cardiac arrest resulting from hanging, drowning, or electrocution will be excluded. Further, patients without a valid personal identification number and non-Danish citizens will be excluded.

Setting The Danish EMS is organised according to the five health regions of Denmark, with an emergency medical dispatch centre in each region. The ground EMS has been supplemented by the Danish Helicopter Emergency Medical Service (HEMS) on a national level since 2014. [14,15] The Danish HEMS is staffed by a consultant-level anaesthesiologist, a pilot and a specially trained paramedic (HEMS crew member).[12] The Danish HEMS is dispatched to time-dependent emergencies such as stroke, cardiac arrest, acute myocardial infarction or severe trauma.[12] The dispatch criteria for the Danish HEMS are described in detail elsewhere. [14,16] The HEMS initiates advanced prehospital interventions both on scene and during transportation; this includes assisted airway management, ultrasound examinations and procedures like thoracotomies and transfusion of blood products. Further, it assures fast transfer to specialised in-hospital care.[14]

Analyses Data will be collected and reported using the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) statement. [17] All data on the personal civil identification number level will be pseudonymised. Descriptive statistics will be reported as absolute numbers and percentages or medians and interquartile ranges. Comparative analyses will be carried out using non-parametric testing to examine subgroups. Normative continuous data will be evaluated with Student's t-test and categorical data with Fisher's exact test. Logistic regression analysis will be performed for multivariate analysis. Due to the low number of survivors, ROSC was chosen as the dependent variable within the adjusted analyses instead of 30-day survival as intended.

The independent association of ROSC will be described using multiple logistic regression with odds ratios (OR) and corresponding (95% CI). The analysis will be adjusted for age, sex, mechanism of injury, response time, initial rhythm and endotracheal intubation. A directed acyclic graph is provided to clarify the basis of the included variables. Statistical significance was considered at a p-value of <0.05, and all statistical tests will be performed using R version 4.1.3 (2022-03-10).

Outcomes The primary outcome is the identification and evaluation of 30-day survival in patients with TCA. The secondary outcomes are the assessment of prehospital ROSC in patients with TCA and status at admission to the hospital. Further, prehospital critical care was evaluated.

Ethical considerations The General Data Protection Regulation will be followed according to Danish legislation, and the study was registered and approved by the Danish Data Protection Agency (Reference: R-22019033 (RS)) and by the Regional Research Board (Reference: REG-031-2022). Since it is a registry-based study, Danish legislation does not require ethical committee approval or patient consent.

Publication The final results are targeted for publication in an international peer-reviewed journal. Participation as coauthors will be decided according to the Vancouver criteria or acknowledged for providing access to data.

ELIGIBILITY:
Inclusion Criteria:

* This study includes all patients (adults and children) with TCA in Denmark between 2016 and 2021 who were treated by the Danish HEMS. Patients will be included if they suffered from an OHCA from traumatic origin and were assessed by the Danish HEMS. The latter will be identified through manual validation based on a predefined search string among all OHCAs in Denmark (derived from the Danish Cardiac Arrest Registry) within the study period.

Exclusion Criteria:

* Patients in whom the HEMS was dispatched but did not arrive will be excluded.
* Patients with cardiac arrest resulting from hanging, drowning, or electrocution will be excluded.
* Further, patients without a valid personal identification number and non-Danish citizens will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises all Danish OHCAs from traumatic origin assessed by the Danish HEMS between 2016 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence pf 30-day survival | 30-Days from incidence.
  30-Days from incidence.

SECONDARY OUTCOMES:
Incidence of prehospital ROSC | Up to 6 hours.
  The incidence of return of spontanous circulation at any time between insult and admission to hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Center, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No